CLINICAL TRIAL: NCT01052103
Title: A 17-Week, Phase 2, Multicenter, Randomized, Double-Blind Study of Treatment With LY2140023 Combined With Standard of Care (SOC) Compared to Placebo With SOC in the Treatment of Patients With Prominent Negative Symptoms of Schizophrenia
Brief Title: A Study of LY2140023 in Schizophrenia Patients With Prominent Negative Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13261; H8Y-MC-HBCO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-13; First posted 2010-01-20 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2140023 (Experimental): 40 mg/day, given orally twice daily (BID) as a 20-mg tablet. LY2140023 dosage was adjustable from 10 mg to 40 mg BID.
  Interventions: Drug: LY2140023; Drug: Standard of Care
- Placebo (Placebo Comparator): Placebo tablets to match LY2140023 tablets
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: LY2140023 — 40 milligrams (mg), oral tablets, twice daily: 20 mg in the morning, 20 mg in the evening, for 16 or 17 weeks. The dose may be adjusted to a minimum of 20 mg or a maximum of 80 mg.
  Other Names: pomaglumetad methionil
  Arms: LY2140023
Drug: Placebo — Placebo oral tablets, twice daily: in the morning and in the evening, for 16 or 17 weeks.
  Arms: Placebo
Drug: Standard of Care — United States (U.S.) label prescribed dose of one of the following Standard of Care Antipsychotics (aripiprazole, olanzapine, risperidone, quetiapine)

SUMMARY:
The purpose of this study is to determine whether LY2140023, when added to standard-of-care antipsychotic treatment, will improve negative symptoms.

DETAILED DESCRIPTION:
The primary objective of this study was to test the hypothesis that treatment with LY2140023 compared to placebo, when added to a fixed dose of a standard of care (SOC) antipsychotic, would demonstrate significantly greater reduction of negative symptoms, as assessed by the 16-item Negative Symptom Assessment scale (NSA-16), in patients with schizophrenia. Patients included in this study were concurrently receiving 1 of 4 second generation antipsychotics (SGAs): aripiprazole, olanzapine, risperidone, or quetiapine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Participants must have been receiving monotherapy treatment for at least 3 months prior to study entry with one of 4 atypical antipsychotic medications (aripiprazole, olanzapine, risperidone, quetiapine)
* Disease symptoms must meet a certain range as assessed by the clinician
* Participants must have evidence of prominent negative symptoms of schizophrenia (for example blunted affect, emotional withdrawal, or motor retardation)
* Participants must be considered reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and be willing to perform all study procedures
* Participants must be able to understand the nature of the study and have given their informed consent

Exclusion Criteria:

* Participants who are actively suicidal
* Participants who are pregnant or nursing
* Participants who have had electroconvulsive therapy (ECT) within 3 months of screening or who will have ECT at any time during the study
* Participants with uncorrected narrow-angle glaucoma, history of or current seizure disorder, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, uncontrolled thyroid condition or other serious or unstable illnesses
* Participants with Parkinson's disease, psychosis related to dementia or related disorders
* Participants with known Human Immunodeficiency Virus positive (HIV+) status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem, Israel
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zamora

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 1-week placebo lead-in period and a 16-week randomization treatment period.
Groups:
- LY2140023 + SOC: 1 week placebo lead-in period followed by 20 milligrams (mg) LY2140023 orally, twice daily for 16 weeks (40 mg/day) treatment period. The dose was allowed to adjust to a minimum of 20 mg/day or a maximum of 80 mg/day plus one of the following Standard of Care (SOC) Antipsychotics (aripiprazole, olanzapine, risperidone, quetiapine) taken per label (United States labeling).
- Placebo + SOC: 1 week placebo lead-in period followed by placebo orally, twice daily for 16 weeks (40 mg/day) plus one of the following SOC Antipsychotics (aripiprazole, olanzapine, risperidone, quetiapine) taken per label (United States labeling) during the treatment period.
Period: Overall Study
Arm/Group | LY2140023 + SOC | Placebo + SOC
Started | 84 | 83
Received at Least 1 Dose of Study Drug | 82 | 82
Completed | 50 | 60
Not Completed | 34 | 23
Not completed — Adverse Event | 10 | 6
Not completed — Entry Criteria Not Met | 3 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Protocol Violation | 10 | 4
Not completed — Scheduling conflict | 2 | 1
Not completed — Sponsor Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Perceived Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2140023 + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.22) | 42.8 (10.23) | 43.3 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 63 | 64 | 127
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black or African American | 41 | 43 | 84
  Multiple | 0 | 2 | 2
  White | 41 | 35 | 76
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 58 | 61 | 119
  Spain | 9 | 7 | 16
  Israel | 11 | 9 | 20
  Italy | 2 | 2 | 4
  Puerto Rico | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 16-Item Negative Symptoms Assessment (NSA-16)
Description: The NSA-16 scale is used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale rates participants on 16 "anchors". Each item ("anchor") is rated from 1 (better) to 6 (worse). The total score is the sum of the 16 specific items and ranges from 16 to 96. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline NSA-16 total score, and baseline NSA-16 total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline NSA-16 total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 81 | 82
units on a scale | -2.7 (1.2) | -3.6 (1.2)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; Changes from baseline to all post-baseline visits were analyzed using a restricted maximum likelihood-based MMRM. Model terms included fixed class effects for visit, investigative site, treatment, SOC type, baseline positive symptom stratum, and treatment-by-visit interaction as well as the continuous, fixed covariates of baseline measurement and baseline-by-visit interaction; Test type: Superiority or Other; p = 0.732, Type 3 Tests — One-sided p-value; LS Mean Differences = 1.0, Standard Error of Mean 1.6

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS Scale consists of 30 items and is designed to measure the severity of psychopathology in schizophrenia. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). The PANSS total score is the sum of the 30 items and has a score ranging from 30 to 210. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline PANSS total score, and baseline PANSS total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline PANSS total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY2140023 + SOC: 1 week placebo lead-in period followed by 20 milligrams (mg) LY2140023, orally, twice daily for 16 weeks (40 mg/day) treatment period. The dose was allowed to adjust to a minimum of 20 mg/day or a maximum of 80 mg/day plus one of the following Standard of Care (SOC) Antipsychotics (aripiprazole, olanzapine, risperidone, quetiapine) taken per label (United States labeling).
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 81 | 82
units on a scale | -4.4 (1.62) | -6.6 (1.55)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.846, Type 3 Tests — One-sided p-value; LS Mean Differences = 2.2, Standard Error of Mean 2.10

3. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale
Description: The CGI-S instrument is used to record the severity of mental illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline CGI-S score, and baseline CGI-S score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline CGI-S measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
units on a scale | -0.4 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.201, Type 3 Tests — One-sided p-value; LS Mean Differences = -0.1, Standard Error of Mean 0.1

4. Secondary Outcome: Change From Baseline in Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery (MCCB) Overall Composite T-Score
Description: MCCB is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The MCCB overall composite T-score combines the individual scores of the 10 tests and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the MCCB overall composite T-score. Higher scores indicate better cognition. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline MCCB overall composite T-score, and baseline MCCB overall composite T-score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline MCCB overall composite T-score measurement.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 58 | 56
T-scores | 3.2 (1.0) | 1.8 (1.0)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.136, Type 3 Tests — One-sided p-value; LS Mean Differences = 1.4, Standard Error of Mean 1.3

5. Secondary Outcome: Change From Baseline in University of California at San Diego Performance-Based Skills Assessment-Brief Version (UPSA-B) Total Score
Description: The UPSA-B is a performance-based assessment of improvement in functional capacity. Participants are asked to role-play tasks in 2 areas of functioning: communication and finances. Raw scores for the 2 subscales are converted into an UPSA-B Total Score (range = 0-100) with higher scores indicating a greater level of functional capacity. Scores of 75 or higher are associated with independent living. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline UPSA-B total score, and baseline UPSA-B total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline UPSA-B total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 62 | 65
units on a scale | 6.5 (1.9) | 4.9 (1.8)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.739, Type 3 Sums of Squares — One-sided p-value; LS Mean Differences = 1.5, Standard Error of Mean 2.4

6. Secondary Outcome: Change From Baseline in Barnes-Akathisia Scale (BAS) Global Score
Description: The BAS is a 4-item instrument that evaluates akathisia associated with use of antipsychotic medications. Item 4 is the Global Clinical Assessment and is rated 0 to 5 (0 = absent, 5 = severe). The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline BAS global score, and baseline BAS global score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline BAS global score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
units on a scale | -0.1 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.190, Type 3 Sums of Squares; LS Mean Differences = -0.1, Standard Error of Mean 0.1

7. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score
Description: The SAS is used to measure Parkinsonian-type symptoms in participants exposed to antipsychotics. SAS consists of 10 items; each rated on a 5-point scale, with 0 meaning complete absence of the condition and 4 meaning the presence of the condition in extreme form. The total score is obtained by adding the ten items, and ranges from 0 to 40. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline SAS total score, and baseline SAS total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline SAS total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
units on a scale | -0.2 (0.2) | -0.1 (0.1)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.702, Type 3 Sums of Squares; LS Mean Differences = -0.1, Standard Error of Mean 0.2

8. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 to 10 are rated on a 5- point scale, with 0 being no dyskinetic movements and 4 being severe dyskinetic movements. Items 11 and 12 are yes/no questions regarding the dental condition of a subject. The AIMS 1-7 total score is the total of items 1 through 7 of the AIMS, and ranges from 0 to 28. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline AIMS 1-7 total score, and baseline AIMS 1-7 total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline AIMS 1-7 total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
units on a scale | 0.0 (0.2) | 0.1 (0.2)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.851, Type 3 Sums of Squares; LS Mean Differences = 0.0, Standard Error of Mean 0.2

9. Secondary Outcome: Number of Participants With Incidence of Epileptiform Activity Outside of Normal Range in Electroencephalograms (EEGs)
Description: Incidence of epileptiform activity outside of normal range in EEGs is based on the changes from normal (E0) or within normal range (E1) at baseline to questionably epileptiform (E2) or clearly epileptiform (E3) or seizure (E4) post-baseline. E0 = Normal; E1 (within normal range) = fewer than 3 focal abnormalities or non-epileptiform abnormalities; E2 (questionably epileptiform) = 3 to 10 focal discharges and/or 1 to 10 multifocal or generalized discharges; E3 (clearly epileptiform) = Sharp/slow complex, runs of epileptiform abnormalities, greater than 10 total epileptiform discharges; and E4 = seizure.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline EEG measurement.
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 80 | 82
participants | 1 | 0

10. Secondary Outcome: Number of Participants With Incidence of Potentially Clinically Significant Changes in Corrected (for Rate) Cardiac QT Interval Using Fridericia's Formula (QTcF) Electrocardiograms (ECGs)
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTcF is the QT interval corrected for heart rate using the Fridericia formula. A potentially clinically significant change in QTcF is defined as >450 milliseconds (ms) for male and >470 ms for female.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline ECG QTcF measurement.
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 81 | 82
participants | 3 | 1

11. Secondary Outcome: Percentage of Participants With a Worsening of Neurological Symptoms From Baseline to Endpoint on the Neurological Examination
Description: Neurological change from baseline was assessed using a 17-item neurological examination and defined as treatment-emergent tremor [increased score on any Item 1- 5; each ranged from 0 (absent) to 3 (interferes with motor function)], nystagmus [increased score for Item 6 or 7; each ranged 0 (absent) to 3 (present on forward gaze)], increased reflexes [increased score and absolute score >2 on any Item 8-11; each ranged 0 (absent) to 4 (clonic)], decreased reflexes [decreased score and absolute score <2 on any Item 8-11; each ranged 0 (absent) to 4 (clonic)], abnormal finger-nose test (Item 12; normal to abnormal), Romberg's sign (Item 13; absent to present), abnormal gait (Item 14; normal to abnormal), decreased muscle strength [decreased score for Item 15 or 16; each ranged 0 (no muscle contraction) to 5 (full and normal power against resistance)], myoclonic jerks [increased score for Item 17; ranged from 0 (absent) to 3 (frequent and across several body regions)].
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline neurological examination.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
percentage of participants
  Tremor | 11.0 | 12.2
  Nystagmus | 2.4 | 2.4
  Increased Reflexes | 3.7 | 4.9
  Decreased Reflexes | 7.3 | 8.5
  Abnormal Finger-Nose Test | 1.2 | 3.7
  Romberg's Sign | 1.2 | 0.0
  Abnormal Gait | 2.4 | 2.4
  Decreased Muscle Strength | 3.7 | 4.9
  Myoclonus Jerks | 4.9 | 2.4

12. Secondary Outcome: Change From Baseline in Standing Blood Pressure (BP)
Description: The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline standing BP, and baseline standing BP*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline standing BP measurement.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
millimeters of mercury (mmHg)
  Standing Systolic BP | -2.0 (1.6) | -2.0 (1.6)
  Standing Diastolic BP | 1.4 (1.1) | -2.4 (1.1)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.999, Type 3 Sums of Squares — P-value is for standing systolic BP; LS Mean Differences = 0.0, 95% CI 2-sided [-4.3 to 4.3]
Statistical Analysis 2: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, Type 3 Sums of Squares — P-value is for standing diastolic BP; LS Mean Differences = 3.8, 95% CI 2-sided [1.0 to 6.7]

13. Secondary Outcome: Change From Baseline in Standing Pulse Rate
Description: The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline standing pulse rate, and baseline standing pulse rate*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline standing pulse rate measurement.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
beats per minute (bpm) | -2.3 (1.7) | -1.8 (1.6)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.818, Type 3 Sums of Squares; LS Mean Differences = -0.5, 95% CI 2-sided [-5.0 to 3.9]

14. Secondary Outcome: Change From Baseline in Weight
Description: The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline weight, and baseline weight*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline weight measurement.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 81 | 81
kilograms (kg) | -1.25 (0.56) | -0.81 (0.55)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.571, Type 3 Sums of Squares; LS Mean Differences = -0.44, 95% CI 2-sided [-1.98 to 1.10]

15. Secondary Outcome: Number of Participants With Incidence of Potentially Clinically Significant (PCS) Change in Laboratory Values Any Time Post-Baseline - General
Description: PCS change in laboratory values were defined as a laboratory value which reached a predefined alert level at any time post-baseline. PCS change in liver function: alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥2* the upper limit of normal (ULN) or total bilirubin ≥1.5*ULN any time post-baseline regardless of the baseline value. Hy's rule: ALT ≥3*ULN, total bilirubin ≥1.5*ULN and alkaline phosphatase <2*ULN at the same time any time post-baseline regardless of the baseline value. PCS change in eosinophil counts: >1.5*10³ cells/microliter any time post-baseline regardless of the baseline value. PCS change in blood creatine phosphokinase: ≥5*ULN any time post-baseline regardless of the baseline value.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug and had at least one post-baseline laboratory measurement.
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
participants
  ALT | 4 | 5
  AST | 1 | 3
  Total bilirubin | 2 | 0
  Hy's rule | 0 | 0
  Eosinophil counts | 0 | 0
  Blood creatine phosphokinase | 7 | 7

16. Secondary Outcome: Number of Participants With Incidence of Potentially Clinically Significant (PCS) Change in Laboratory Values Any Time Post-Baseline - Fasting Cholesterol
Description: PCS change in laboratory values were defined as a laboratory value which reached a predefined alert level at any time post-baseline. PCS change in total cholesterol: Normal (N) to High (H) <200 milligrams/deciliter (mg/dL) at baseline and ≥240 mg/dL post-baseline; Borderline (B) to H ≥200 mg/dL and <240 mg/dL at baseline and ≥240 mg/dL post-baseline; N/B to H <240 mg/dL at baseline and ≥240 mg/dL post-baseline; N to B/H <200 mg/dL at baseline, ≥200 mg/dL post-baseline. PCS change in low-density lipoprotein (LDL) cholesterol: N to H <100 mg/dL at baseline and ≥160 mg/dL post-baseline; B to H ≥100 mg/dL and <160 mg/dL at baseline and ≥160 mg/dL post-baseline; N/B to H <160 mg/dL at baseline and ≥160 mg/dL post-baseline; N to B/H <100 mg/dL at baseline, ≥100 mg/dL post-baseline. PCS change in high-density lipoprotein (HDL) cholesterol: ≥40 mg/dL at baseline and <40 mg/dL post-baseline.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had normal or borderline cholesterol level at baseline and at least one post-baseline cholesterol measurement. "Number" represents number of participants with an incidence of potentially clinically significant (PCS) change in laboratory values
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 73 | 68
participants
  Total Cholesterol N to H: number analyzed (Participants) | 35 | 42
  Total Cholesterol N to H | 1 | 0
  Total Cholesterol B to H: number analyzed (Participants) | 36 | 25
  Total Cholesterol B to H | 8 | 7
  Total Cholesterol N/B to H: number analyzed (Participants) | 71 | 67
  Total Cholesterol N/B to H | 9 | 7
  Total Cholesterol N to B/H: number analyzed (Participants) | 35 | 42
  Total Cholesterol N to B/H | 9 | 9
  LDL Cholesterol N to H: number analyzed (Participants) | 22 | 13
  LDL Cholesterol N to H | 0 | 0
  LDL Cholesterol B to H: number analyzed (Participants) | 42 | 55
  LDL Cholesterol B to H | 13 | 13
  LDL Cholesterol N/B to H: number analyzed (Participants) | 64 | 68
  LDL Cholesterol N/B to H | 13 | 13
  LDL Cholesterol N to B/H: number analyzed (Participants) | 22 | 13
  LDL Cholesterol N to B/H | 9 | 2
  HDL Cholesterol N to Low: number analyzed (Participants) | 73 | 66
  HDL Cholesterol N to Low | 24 | 24

17. Secondary Outcome: Number of Participants With Incidence of Potentially Clinically Significant (PCS) Change in Laboratory Values Any Time Post-Baseline - Fasting Triglycerides
Description: PCS change in laboratory values were defined as a laboratory value which reached a predefined alert level at any time post-baseline. PCS change for Normal (N) to High (H) <150 milligrams/deciliter (mg/dL) at baseline and ≥200 mg/dL post-baseline; N/Borderline (B) to H <200 mg/dL at baseline and ≥200 mg/dL post-baseline; N to very H <150 mg/dL at baseline and ≥500 mg/dL post-baseline; B to H >150 and <200 mg/dL at baseline and ≥200 mg/dL post-baseline; B to very H >150 and <200 mg/dL at baseline and ≥500 mg/dL post-baseline; N/B to very H <200 mg/dL at baseline and ≥500 mg/dL post-baseline; N to B/H/very H <150 mg/dL at baseline and ≥150 mg/dL post-baseline.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had normal or borderline triglycerides level at baseline and at least one post-baseline triglycerides measurement. "Number" represents number of participants with an incidence of potentially clinically significant (PCS) change in laboratory values
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 67 | 59
participants
  N to H: number analyzed (Participants) | 51 | 45
  N to H | 10 | 7
  N/B to H | 20 | 13
  N to very H: number analyzed (Participants) | 51 | 45
  N to very H | 0 | 0
  B to H: number analyzed (Participants) | 16 | 14
  B to H | 10 | 6
  B to very H: number analyzed (Participants) | 16 | 14
  B to very H | 0 | 0
  N/B to very H | 0 | 0
  N to B/H/very H: number analyzed (Participants) | 51 | 45
  N to B/H/very H | 18 | 17

18. Secondary Outcome: Number of Participants With Incidence of Potentially Clinically Significant (PCS) Change in Laboratory Values Any Time Post-Baseline - Fasting Glucose
Description: PCS change in laboratory values were defined as a laboratory value which reached a predefined alert level at any time post-baseline. PCS change for Normal to High: <100 milligrams/deciliter (mg/dL) at baseline and ≥126 mg/dL post-baseline; Impaired to High ≥100 mg/dL and <126 mg/dL at baseline and ≥126 mg/dL any time post-baseline; Normal/Impaired to High <126 mg/dL at baseline and ≥126 mg/dL any time post-baseline.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had normal or impaired glucose level at baseline and at least 1 post-baseline glucose measurement. "Number" represents number of participants with an incidence of potentially clinically significant (PCS) change in laboratory values
Measure: Number; unit: participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 74 | 76
participants
  Normal to High: number analyzed (Participants) | 39 | 46
  Normal to High | 2 | 8
  Impaired to High: number analyzed (Participants) | 35 | 30
  Impaired to High | 10 | 5
  Normal/Impaired to High | 12 | 13

19. Secondary Outcome: Percentage of Participants With Incidence of Potentially Clinically Significant Change of Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Percentage of participants with incidence of potentially clinically significant change of the C-SSRS was calculated as the number of participants with an increase in suicidal behavior or ideation over baseline, divided by the total number of participants multiplied by 100.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline C-SSRS measurement.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
percentage of participants
  Treatment-Emergent Suicidal Ideation | 2.4 | 4.9
  Treatment-Emergent Suicidal Behavior | 0.0 | 1.2
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.682, Fisher Exact — P-value is for treatment-emergent suicidal ideation

20. Secondary Outcome: Change From Baseline to Endpoint in Personal and Social Performance (PSP) Scale
Description: The PSP scale is a 100-point, single item, clinician-rated scale to assess a participant's overall functioning, including personal and social relationships, socially useful activities, self-care, and disturbing and aggressive behaviors. The higher scores indicate a higher level of functioning. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline PSP score, and baseline PSP score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline PSP measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 75 | 77
units on a scale | 8.9 (1.3) | 7.9 (1.3)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.727, Type 3 Sums of Squares — One-sided p-value; LS Mean Differences = 1.0, Standard Error of Mean 1.7

21. Secondary Outcome: Time to Discontinuation From the Study Due to Any Reason
Description: The time to discontinuation due to any reason was defined as the total number of days between the date of first dose and discontinuation date. The time to discontinuation was analyzed using Kaplan-Meier estimated survival curves. Participants who completed the study were considered censored. Less than 50% of participants discontinued from study at randomization treatment Week 16 endpoint, therefore median values were not calculated.
Time Frame: First dose to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug. Participants who completed the study were considered censored: 50 for LY2140023 + SOC group and 60 for placebo + SOC group.
Measure: Median (Full Range); unit: months
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 82 | 82
months | NA [NA to NA] — The median (full range) was not calculated because an insufficient number of participants reached the event at the final time point (randomization treatment Week 16). | NA [NA to NA] — The median (full range) was not calculated because an insufficient number of participants reached the event at the final time point (randomization treatment Week 16).

22. Secondary Outcome: Schizophrenia Resource Use Module (S-RUM) - Number of Emergency Room (ER) or Equivalent Facility Visits and Outpatient Medical Visits
Description: The S-RUM is a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, ER visits, and outpatient medical visits for a specified period of time. Item 1 asks about the number of ER or equivalent facility visits a participant had for psychiatric (psych) illness. Item 2 asks about the number of ER or equivalent facility visits a participant had for non-psychiatric (non-psych) illness or injury. Item 5 asks about the number of outpatient visits to other physicians (not psychiatrists or dentists).
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug and had S-RUM assessment.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 80 | 80
visits
  ER/Facility (Psych) visits | 0.6 (4.11) | 0.2 (1.79)
  ER/Facility (Non-Psych) visits | 0.2 (0.43) | 0.1 (0.56)
  Outpatient (Non-Psych or Dentist) visits | 0.7 (1.33) | 1.2 (2.99)

23. Secondary Outcome: Schizophrenia Resource Use Module (S-RUM) - Number of Sessions With a Psychiatrist
Description: The S-RUM is a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, Emergency Room (ER) visits, and outpatient medical visits for a specified period of time. Item 4 asks about the number of sessions with a psychiatrist a participant had.
Time Frame: Baseline to randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug and had S-RUM assessment.
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 80 | 80
sessions | 3.4 (17.49) | 1.5 (2.76)

24. Secondary Outcome: Change From Baseline to Endpoint in the EuroQol Questionnaire-5 Dimension (EQ-5D) Visual Analog Scale (VAS) Health State Score
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument that contains 2 parts: a health status profile and a visual analog scale (VAS) to rate global health-related quality of life. VAS health state scores range from 0 (worst imaginable health state) to 100 (best imaginable health state). The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline VAS health state score, and baseline VAS health state score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline VAS health state measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 74 | 77
units on a scale | 3.7 (2.6) | 5.4 (2.4)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.305, Type 3 Sums of Squares — One-sided p-value; LS Mean Differences = -1.7, Standard Error of Mean 3.4

25. Secondary Outcome: Change From Baseline to Endpoint in the Subjective Well-Being Under Neuroleptic Treatment-Short Form (SWN-SF) Total Score
Description: The SWN-SF measures subjective well-being for the previous 7 days. The 20-item scale covers 5 health domains (subscales; 4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). Each of the 5 subscale scores range from 4 to 24. SWN-SF total scores range from 20 to 120. Higher scores indicate greater well-being. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for visit, pooled investigative site, treatment, standard of care (SOC) type, baseline positive symptom stratum, treatment*visit, baseline SWN-SF total score, and baseline SWN-SF total score*visit.
Time Frame: Baseline, randomization treatment Week 16
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline SWN-SF total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023 + SOC | Placebo + SOC
Number analyzed (Participants) | 73 | 75
units on a scale | 3.9 (2.0) | 4.4 (1.9)
Statistical Analysis 1: Comparison: LY2140023 + SOC vs Placebo + SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.420, Type 3 Sums of Squares — One-sided p-value; LS Mean Differences = -0.5, Standard Error of Mean 2.5

ADVERSE EVENTS:
Arm/Group | LY2140023 + SOC | Placebo + SOC
Serious Adverse Events (participants affected / at risk) | 8/82 | 4/82
Other Adverse Events (participants affected / at risk) | 54/82 | 51/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2140023 + SOC (N=82) | Placebo + SOC (N=82)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 3 (3) | 1 (1)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2140023 + SOC (N=82) | Placebo + SOC (N=82)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 9 (9)
Nausea (Gastrointestinal disorders) | 11 (12) | 4 (4)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (13) | 2 (7)
Fatigue (General disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 1/19 (1) | 0/18 (0)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 7 (7)
Weight increased (Investigations) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Akathisia (Nervous system disorders) | 1 (1) | 4 (5)
Dizziness (Nervous system disorders) | 3 (4) | 3 (3)
Headache (Nervous system disorders) | 11 (12) | 11 (12)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days